CLINICAL TRIAL: NCT03906513
Title: Evaluation of the Efficacy of OMK2 in Recovering Corneal Neural Damage in Patients With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Paolo Fogagnolo, Researcher, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OMK20915
Record Dates: First submitted 2019-04-04; First posted 2019-04-08 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Cornea
Keywords: Cornea; Diabetes; Neural damage
MeSH Terms: conditions — Corneal Diseases; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Active Comparator): 20 patients will be treated with active treatment (OMK2)
  Interventions: Device: OMK2
- Placebo (Placebo Comparator): 10 patients will be treated with placebo (lubricant eye drops)
  Interventions: Device: OMK2

INTERVENTIONS:
Device: OMK2 — OMK2 (including citicoline 2%, high molecular weight hyaluronic acid 0.2%, cyanocobalamin and 0.01% BAK, Omikron Italia SRL) is a Class IIa device CE marked registered in Medical Devices Database of Italian Ministry of Health (identification number of registration: 1170558).

SUMMARY:
This will be a single-centre, randomized, pilot study. 30 patients with diabetes who previously had received Argon laser photocoagulation will be enrolled.

DETAILED DESCRIPTION:
This will be a single-centre, randomized, pilot study. 30 patients with diabetes who previously had received Argon laser photocoagulation will be enrolled. These patients will receive corneal esthesiometry and will be divided in those with esthesiometry < 45 mm [6] (clinically detectable corneal neuropathy, CDCN) and not (NCDCN).

Patients will be randomized to the two treatment arms: 20 patients will be treated with active treatment (OMK2) and 10 patients will be treated with placebo (lubricant eye drops) given three times daily (8 am, 2 pm, 8 pm) for 18 months. Stratification for (1) CDCN, (2) duration of the disease, and (3) insulin-dependent diabetes will be adopted.

The randomization will be operator-masked.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Type 1 or type 2 diabetic patients who received Argon Laser Photocoagulation

Exclusion Criteria:

* Neuropathy of any other cause than diabetes
* A history of conditions known to affect corneal sensitivity
* Coexisting other corneal diseases
* Autoimmune diseases
* Sjogren syndrome
* History of corneal trauma
* Contact lenses users
* Patients needing eye surgery or who received eye surgery at least 180 days before study beginning.
* contraindications to the use of any active substances and/or excipients
* pregnant and lactating women
* pediatric patients or adolescents under 18 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2017-05-03 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
changes in the characteristics of the subbasal corneal plexus at confocal | Change measure (baseline and month 18)
  changes in the characteristics of the subbasal corneal plexus at confocal microscopy (central + 8 paracentral quadrants)
  * changes in corneal esthesiometry (Cochet-Bonnet esthesiometer); central and four quadrants changes in the characteristics of the subbasal corneal plexus at confocal microscopy (central + 8 paracentral quadrants)
  * changes in corneal esthesiometry (Cochet-Bonnet esthesiometer); central and changes in the characteristics of the subbasal corneal plexus at confocal microscopy (central + 8 paracentral quadrants)
  * changes in corneal esthesiometry (Cochet-Bonnet esthesiometer); central and four quadrants four quadrants

SECONDARY OUTCOMES:
- changes in clinical signs and symptoms of ocular surface damage | Change measure (baseline and month 18)
  * changes in clinical signs of corneal damage (BUT, Schirmer I, corneal and conjunctival epithelial staining using Oxford and Van Bijelsterveld scales, both ranging between 0 - normal, to 4 - severely affected; a change of 1 or more stage is defined as clinically relevant)
  * changes in symptoms (OSDI)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Fogagnolo, MD, Principal Investigator — University of Milan
Locations (1):
- ASST Santi Paolo e Carlo - Ospedale San Paolo, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fogagnolo P, Melardi E, Tranchina L, Rossetti L. Topical citicoline and vitamin B12 versus placebo in the treatment of diabetes-related corneal nerve damage: a randomized double-blind controlled trial. BMC Ophthalmol. 2020 Aug 1;20(1):315. doi: 10.1186/s12886-020-01584-w. PMID 32738875